CLINICAL TRIAL: NCT02599545
Title: Testosterone and Cortisol Levels in Infant Health and Development
Brief Title: Testosterone and Cortisol Levels in Infants
Status: Terminated | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00065480
Record Dates: First submitted 2015-10-29; First posted 2015-11-06 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2017-07

CONDITIONS: Infant, Premature; Infant, Very Low Birth Weight
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be obtained only from the infant by collecting the leftover cord blood from the hospital lab. If no remnant blood is available, a blood specimen will not be collected. Mothers will be asked to provide a saliva sample within 72 hours of delivery, then mother and infant saliva sampling will be collected in the morning on the same day when the infant reaches 40 weeks postmenstrual age (PMA) or discharge from the Duke Intensive Care Nursery (ICN) (whichever comes first), 12 months, and 24 months corrected age (CA)(+/- 1 month).

GROUPS / COHORTS (1):
- Maternal/VLBW Infant Pairs: One-hundred-fifty mother-VLBW infant pairs, a total of 300 participants, will be recruited for the final sample size of 120 pairs.

SUMMARY:
Very low birth weight (VLBW) infants have more health and developmental problems than normal birth weight full-term infants. These problems are more common in males than female VLBW preterm infants. Male VLBW infants also experience less positive mother-infant interactions than females, especially when mothers are emotionally distressed. This is a significant problem because positive mother-infant interactions function as an important protective factor against the negative health and developmental outcomes associated with prematurity. The source of the vulnerability of male VLBW infants to health problems, suboptimal mother-infant interactions, and poor development goes beyond gender socialization differences and includes biological factors. Identification of infant and maternal biological markers/predictors of infant health and developmental outcomes could ultimately lead to interventions for VLBW preterm infants.

The purpose of this study is to confirm that testosterone rather than cortisol is a more reliable marker/predictor of complications affecting infants' health outcomes, mother-infant interactions, and infant cognitive/motor/language developmental outcomes; and that male infants exhibit a higher sensitivity to testosterone levels than female infants.

This longitudinal study will examine the associations of the steroid hormones, testosterone and cortisol, levels with infant health, mother-infant interactions, and infant cognitive/motor/language development ('infant development') in very low birthweight (VLBW, BW < 1,500 g) preterm (gestational age < 32 weeks gestation) infants after adjusting for maternal physical and mental health state, infant socioemotional and behavioral development, and characteristics of infants and mothers. Concurrent and repeated measurement of testosterone and cortisol levels both in infants and mothers will be conducted through infancy and early childhood (at birth, 40 weeks postmenstrual age, 12 and 24 months corrected age).

ELIGIBILITY:
Inclusion Criteria:

* Neonates will be included if they are less than or equal to 32/0 weeks gestational age at birth and have a birth weight < 1500 grams.
* Mothers will be included if they are (1) older than 15 years, (2) able to communicate in English or Spanish, (3) primary caregivers of the newborn.

Exclusion Criteria:

* Neonates will be excluded if they (1) are born > 32/0 weeks GA, (2) weigh more than 1,500 grams at birth, (3) have congenital abnormalities, (2) will be discharged before day 7 of life, (3) have a positive urine drug screen, or (4) are being placed for adoption after discharge from the hospital.
* Mothers will be excluded if they have (1) narcotic or injection drug dependence or (2) a documented serious health (e.g., cancer or HIV positive) or psychological (e.g., schizophrenia) problem.

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mothers will be eligible for consent if they are a patient in the Duke University Hospital Labor & Delivery department and meet all eligibility criteria. Potential mothers will be approached about the study before delivery or within 72 hours after delivery. 150 mother-VLBW infant pairs, a total of 300 participants, will be recruited for the final sample size of 120 pairs. English or Spanish speaking mothers may participate. If the mother is between 15-17 years of age, a minor mother consent will be used. If the mother is Spanish speaking, a Spanish short form consent will be used with a Spanish interpreter. If the mother is pre-consented, the infant may or may not be enrolled at delivery. The infant could be excluded if he/she is delivered at a gestation or weight that is outside of study limits, or if she/he has a severe health problem/congenital anomaly detected at birth.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
measurements of maternal and neonate/infant testosterone and cortisol (T&C) levels from admission through 24-months of life to determine associations of T&C with health outcomes of neonates and infants between genders | Admission through 24 months of life
  The levels of testosterone and cortisol will be measured and compared with health outcomes of neonates/infants, at birth, 40 weeks postmenstrual age (PMA), 6, 12, and 24 months corrected age (CA) after controlling for covariates. The latter include maternal psychological state, infant temperament, and characteristics of mothers (age, race, body mass index [BMI], education, and marital status).
video recorded interactions at 12- and 24-months to determine associations of testosterone and cortisol levels with quality of mother-infant interactions between genders during infancy | 12- and 24-months of age
  The levels of testosterone and cortisol will be measured and compared with quality of mother-infant interactions at 12- and 24-months CA after controlling for the covariates.
standard infant testing at 12- and 24-months of age to determine associations of testosterone and cortisol levels with infant cognitive/motor/language development between genders during infancy | 12- and 24-months of age
  The levels of testosterone and cortisol will be measured and compared with infant development at 12- and 24-months CA after controlling for the covariates and mother-infant interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. June Cho, PhD, RN, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States